CLINICAL TRIAL: NCT05731479
Title: Effectiveness of a Radiofrequency Diathermy and Therapeutic Exercise Protocol in Women With Abdominal Diastasis. Randomized Controlled Trial
Brief Title: Radiofrequency Diathermy and Therapeutic Exercise Protocol in Women With Abdominal Diastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2524988
Record Dates: First submitted 2023-01-26; First posted 2023-02-16 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-12

CONDITIONS: Abdominal Diastasis
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diathermy + exercise group (Experimental): Application of diathermy and a therapeutic exercise protocol.
  Interventions: Other: Diathermy + exercise group
- Diathermy placebo + exercise group (Placebo Comparator): Application of the diathermy device without energy emission and a therapeutic exercise protocol.
  Interventions: Other: Diathermy placebo + exercise group

INTERVENTIONS:
Other: Diathermy + exercise group — The Diathermy + Exercise group will receive diathermy for 15 minutes, of which 5 minutes will be applied in the capacitive method and 10 minutes in the resistive method. You will then perform 20 minutes of the following exercises: 1) Bird-Dog, 2) Crunch, 3) Obliques, 4) Drawing, 5) Half plank and 6) Side-plank. You will perform 8-12 repetitions and 3 sets of each exercise. 3 sessions of 35 minutes per week for 8 weeks.
  Arms: Diathermy + exercise group
Other: Diathermy placebo + exercise group — The Placebo + Exercise group will receive 15 minutes of application of the diathermy device without energy emission. It will then perform the same therapeutic exercise protocol described in the GDE. 3 sessions of 35 minutes per week for 8 weeks.
  Arms: Diathermy placebo + exercise group

SUMMARY:
Diastasis recti abdominis (DRA) is defined as the presence of divergence between the rectus abdominis muscles along the linea alba. DRA is associated with decreased abdominal strength and degraded health and physical functioning, which results in poorer body perception and satisfaction and negatively affects the quality of life in its multiple spheres (social, sexual and personal). Regarding the different treatment techniques for DRA, different treatments have been described, such as bandages, electrotherapy or therapeutic exercise, the latter being the most scientifically supported option to approach DRA conservatively. Exercise has shown positive effects on DRA severity, abdominal muscle thickness, abdominal strength and endurance, and quality of life in women with DRA.

Another treatment that has shown promising effects in various pathologies is radiofrequency diathermy using the Capacitive-Resistive Electrical Transfer system. The capacitive mode acts on soft tissues containing electrolytes such as muscles and vascular and lymphatic tissues. On the other hand, the resistive mode acts on tissues of higher density and fat and fiber content, such as bones, ligaments and tendons. It has been documented that this type of therapy acts favoring the vascularization of tissues, decreasing inflammation and favoring the processes of cellular repair and analgesia. Its beneficial effect on low back pain and various pelvic floor disorders has been studied. However, at present, there are no studies evaluating the effectiveness of this type of intervention in people with abdominal diastasis.

In view of the above, the objective of our study is to evaluate the effectiveness of a protocol based on therapeutic exercise preceded by a radiofrequency diathermy program on anthropometric parameters, anatomo-physiological parameters, functional parameters, and parameters related to psychological aspects in women with postpartum abdominal diastasis.

DETAILED DESCRIPTION:
A longitudinal randomized controlled experimental study will be carried out. The sample will be composed of 34 postpartum women, randomly distributed in two groups: i) diathermy + exercise group (GDE) (n=17), and ii) placebo diathermy + exercise group (GPE) (n=17).

The evaluations will be performed at two time points: i) before the intervention (T1), and ii) after the last session (T2).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45 years,
* 3 to 24 months postpartum
* Criteria of abdominal diastasis according to Beer's criteria (Beer et al.2009)

Exclusion Criteria:

* Rejection to sign the informed consent form
* Presence of any metabolic, neurological or connective tissue disease, as well as cognitive alterations.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rectus abdominis distance | Baseline
  The distance between rectus abdominis in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Rectus abdominis distance | Immediately after the intervention
  The distance between rectus abdominis in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Rectus abdominis thickness | Baseline
  The rectus abdominis thickness in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Rectus abdominis thickness | Immediately after the intervention
  The rectus abdominis thickness in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.

SECONDARY OUTCOMES:
Body composition | Baseline
  Body composition by means of Bioimpedance (Tanita DC-430MA, Tanita Corporation of America, Inc., Arlington Heights, IL, USA).
Body composition | Immediately after the intervention
  Body composition by means of Bioimpedance (Tanita DC-430MA, Tanita Corporation of America, Inc., Arlington Heights, IL, USA).
Strength of the abdominal flexor musculature | Baseline
  Strength of the abdominal flexor musculature by means of a dynamometer (Lafayette, Indiana, USA)
Strength of the abdominal flexor musculature | Immediately after the intervention
  Strength of the abdominal flexor musculature by means of a dynamometer (Lafayette, Indiana, USA)
Kinesiophobia | Baseline
  Kinesiophobia with the Tampa Scale of Kinesiophobia-11 questionnaire: It maintains items 1, 2, 3, 5, 6, 7, 10, 11, 13, 15, and 17 from the original 17-point scale, and its score ranges from 11-44, where the lowest 11 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Kinesiophobia | Immediately after the intervention
  Kinesiophobia with the Tampa Scale of Kinesiophobia-11 questionnaire: It maintains items 1, 2, 3, 5, 6, 7, 10, 11, 13, 15, and 17 from the original 17-point scale, and its score ranges from 11-44, where the lowest 11 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia
Body image | Baseline
  Body image using the Multidimensional Body Self Relations Questionnaire: It consists of 69 items each rated on a 5-point scale from 1 to 5 (strongly disagree-strongly agree). The higher the score, the greater the satisfaction with one's own body image, so the total score of the instrument requires reversing the score of the items that indicate dissatisfaction
Body image | Immediately after the intervention
  Body image using the Multidimensional Body Self Relations Questionnaire: It consists of 69 items each rated on a 5-point scale from 1 to 5 (strongly disagree-strongly agree). The higher the score, the greater the satisfaction with one's own body image, so the total score of the instrument requires reversing the score of the items that indicate dissatisfaction
Perception of change after the intervention | Baseline
  Perception of change after the intervention with the Patient Perception of Change after Treatment questionnaire. consisting of a verbal scale, with 7 points "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", "very much worse".
Perception of change after the intervention | Immediately after the intervention
  Perception of change after the intervention with the Patient Perception of Change after Treatment questionnaire. consisting of a verbal scale, with 7 points "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", "very much worse".
Linea alba thickness | Baseline
  Linea alba thickness in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Linea alba thickness | Immediately after the intervention
  Linea alba thickness in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Linea alba distortion index | Baseline
  Linea alba distortion index in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Linea alba distortion index | Immediately after the intervention
  Linea alba distortion index in millimetres (mm) will be assessed with an ultrasound machine, using a high-resolution linear array transducer.
Stabilization capacity and resistance of the abdomino-lumbo-pelvic capsule | Baseline
  Stabilization capacity and resistance of the abdomino-lumbo-pelvic capsule, with a battery of validated maneuvers: gluteal bridge, gluteal bridge with unipodal support, lateral planks and horizontal plank.
  The measurement unit is the second (s) for all maneuvers, and the time for each manoeuvre shall be averaged.
Stabilization capacity and resistance of the abdomino-lumbo-pelvic capsule | Immediately after the intervention
  Stabilization capacity and resistance of the abdomino-lumbo-pelvic capsule, with a battery of validated maneuvers: gluteal bridge, gluteal bridge with unipodal support, lateral planks and horizontal plank.
  The measurement unit is the second (s) for all maneuvers, and the time for each manoeuvre shall be averaged.
Abdominal circumference | Baseline
  Abdominal circumference will be assessed by means of tape measure in centimetres (cm). Two measurements shall be taken and averaged.
Abdominal circumference | Immediately after the intervention
  Abdominal circumference will be assessed by means of tape measure in centimetres (cm). Two measurements shall be taken and averaged.
Abdominal fold | Baseline
  Abdominal fold will be assessed by means of a plicometer in milimetres (mm). Two measurements shall be taken and averaged.
Abdominal fold | Immediately after the intervention
  Abdominal fold will be assessed by means of a plicometer in milimetres (mm). Two measurements shall be taken and averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Inglés, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gluppe SB, Engh ME, Bo K. Immediate Effect of Abdominal and Pelvic Floor Muscle Exercises on Interrecti Distance in Women With Diastasis Recti Abdominis Who Were Parous. Phys Ther. 2020 Aug 12;100(8):1372-1383. doi: 10.1093/ptj/pzaa070. PMID 32302393
- [Background] Keshwani N, Mathur S, McLean L. The impact of exercise therapy and abdominal binding in the management of diastasis recti abdominis in the early post-partum period: a pilot randomized controlled trial. Physiother Theory Pract. 2021 Sep;37(9):1018-1033. doi: 10.1080/09593985.2019.1675207. Epub 2019 Oct 23. PMID 31642725
- [Background] Thabet AA, Alshehri MA. Efficacy of deep core stability exercise program in postpartum women with diastasis recti abdominis: a randomised controlled trial. J Musculoskelet Neuronal Interact. 2019 Mar 1;19(1):62-68. PMID 30839304